CLINICAL TRIAL: NCT00201825
Title: A Phase II Study of Capecitabine and Docetaxel in Previously Untreated Advanced Non-Small Cell Lung Cancer Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tony Bekaii-Saab (Other)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Sponsor-Investigator, Tony Bekaii-Saab, Principal Investigator, Ohio State University Comprehensive Cancer Center
Organization: Ohio State University Comprehensive Cancer Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSU-0356; NCI-2011-03593 (Registry Identifier: CTRP (Clinical Trials Reporting Program))
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Results first posted 2014-10-06 (Estimated); Last update posted 2014-10-06 (Estimated); Status verified 2014-10

CONDITIONS: Lung Cancer; Non-Small-Cell Lung Carcinoma
Keywords: Previously Untreated; Advanced
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Capecitabine; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Docetaxel and Capecitabine (Experimental)
  Interventions: Drug: Capecitabine; Drug: Docetaxel

INTERVENTIONS:
Drug: Capecitabine — 1250 mg/m2/day in 2 oral daily divided doses of 625 mg/m2 on day 5 of every cycle and continued for 14 days.
  Other Names: Xeloda
Drug: Docetaxel — 36 mg/m2 IV weekly for 3 weeks every 4 weeks.
  Other Names: Taxotere

SUMMARY:
This study will determine the objective response rate in chemotherapy naive non-small cell lung cancer patients with advanced disease.

DETAILED DESCRIPTION:
Rationale: Docetaxel has some efficacy against non-small cell lung cancer (NSCLC). This drug is Food and Drug Administration approved in combination with cisplatin (Platinol) for the treatment of unresectable, locally advanced or metastatic NSCLC in patients who have not previously had chemotherapy for this condition. Docetaxel is also approved for second line treatment of metastatic NSCLC. Research indicates that capecitabine, in combination with docetaxel, has efficacy against NSCLC. Capecitabine appears to have anti-cancer activity through several enzymes. This drug is metabolized in the body to another agent called 5-FU. During this conversion process, 5-FU requires thymidine phosphorylase (TP), a cellular characteristic associated with tumor growth. There are higher levels of TP expression in tumors as compared to normal tissue. The drug administration schedule in this study is designed to optimize efficacy against the TP target through both docetaxel and capecitabine. This study will measure biological changes to TP and other enzymes to help researchers gain more information about how capecitabine and docetaxel works against NSCLC.

Purpose: This study will evaluate the efficacy of docetaxel and capecitabine in patients with previously untreated advanced NSCLC. Tests related to tumor biology will be conducted before and during study treatments and correlated with patient responses to therapies.

Treatment: Patients in this study will receive docetaxel and capecitabine. Docetaxel will be administered through intravenous infusions. Capecitabine will be provided through oral pills. A four-week period constitutes one cycle. Docetaxel will be given weekly for three weeks followed by one week of rest. Capecitabine will be taken twice daily on days 5 through 14 of the treatment cycle. Several tests and exams will be given throughout the study to closely monitor patients. Treatments will be discontinued due to disease growth or unacceptable side effects.

ELIGIBILITY:
Inclusion Criteria:

* Must have advanced NSCLC
* No prior chemotherapy
* Eastern Cooperative Oncology Group(ECOG)Performance Status:0 or 1
* Must have measurable disease (RECIST criteria)
* life expectancy of at least 12 weeks
* adequate organ function including

Exclusion Criteria:

* Pregnant or lactating women
* Psychiatric disorders that would interfere w/consent or follow-up
* Patients with uncontrolled diabetes mellitus, defined as random blood sugar > 250mg/dL.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2004-12; Primary Completion 2012-12 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tony Bekaii-Saab, Principal Investigator — Ohio State University
Locations (1):
- Ohio State University, Columbus, Ohio, United States

REFERENCES:
- [Result] Bertino EM, Bekaii-Saab T, Fernandez S, Diasio RB, Karim NA, Otterson GA, Villalona-Calero MA. A phase II study of modulated-capecitabine and docetaxel in chemonaive patients with advanced non-small cell lung cancer (NSCLC). Lung Cancer. 2013 Jan;79(1):27-32. doi: 10.1016/j.lungcan.2012.09.013. Epub 2012 Oct 16. PMID 23079156
- See also: Jamesline — http://cancer.osu.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were enrolled and received treatment between December 2004 and November 2007
Period: Overall Study
Arm/Group | Docetaxel and Capecitabine
Started | 29
Completed | 29
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Eligible patients had histologically confirmed advanced NSCLC and had not received prior chemotherapy.
Arm/Group | Docetaxel and Capecitabine
Number analyzed (Participants) | 29
Age, Continuous [Median (Full Range); unit: years] | 61 [39 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 22
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 25
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: patients]
  United States | 29
Histology [Number; unit: patients]
  Adenocarcinoma | 13
  Squamous cell carcinoma | 6
  Large cell Carcinoma | 2
  NSCLC not specified | 8
ECOG (Eastern Cooperative Oncology Group) [Number; unit: patients]
  Performance status 0 (Fully active) | 8
  Performance status 1 (Restricted activity) | 21

OUTCOME MEASURES:

1. Primary Outcome: Determine Objective Response Rate
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: Every 35 days
Population: One patient was not evaluable for response because the patient was removed from study afer an adverse event.
Measure: Number; unit: patients
Arm/Group | Docetaxel and Capecitabine
Number analyzed (Participants) | 28
patients
  Complete response (CR) | 0
  Partial response (PR) | 5
  Stable Disease | 14
  Disease Progression | 9
  Overall response (CR + PR) | 5

2. Secondary Outcome: Time to Tumor Progression
Time Frame: Every 35 days
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Docetaxel and Capecitabine
Number analyzed (Participants) | 28
months | 3.3 [1.5 to 4.6]

3. Secondary Outcome: One Year Survival
Time Frame: one year
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Docetaxel and Capecitabine
Number analyzed (Participants) | 28
months | 10.5 [3.2 to 15]

4. Secondary Outcome: Pharmacokinetics
Time Frame: Cycle 2
Population: No Pharmacokinetics were conducted for this trial.
Arm/Group | Docetaxel and Capecitabine
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse events were assessed using the NCI Common Toxicity Criteria version 3.0 from week 1 of the study until end of study.
Description: Adverse events will use the descriptions and grading scales found in the revised NCI Common Toxicity Criteria (CTC). This study will utilize the CTC version 3.0 for toxicity and Adverse Drug Experience reporting.
Arm/Group | Docetaxel and Capecitabine
Serious Adverse Events (participants affected / at risk) | 1/29
Other Adverse Events (participants affected / at risk) | 29/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Docetaxel and Capecitabine (N=29)
Myocardial infarction (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Docetaxel and Capecitabine (N=29)
Anemia (Blood and lymphatic system disorders) | 15 (15)
Neutropenia (General disorders) | 10 (10)
Leukopenia (Investigations) | 21 (21)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No